CLINICAL TRIAL: NCT03336359
Title: Tandem Colonoscopy Study of Linked Color Imaging Versus Narrow Band Imaging on Colorectal Adenoma Detection: A Prospective, Randomized Study
Brief Title: Linked Color Imaging Versus Narrow Band Imaging for Colorectal Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LINA
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Colon Adenoma
Keywords: colonoscopy; image enhanced endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCI (Active Comparator): Tandem colonoscopy with Linked Color Imaging system
  Interventions: Diagnostic Test: Tandem colonoscopy
- NBI (Active Comparator): Tandem colonoscopy with Narrow band imaging system
  Interventions: Diagnostic Test: Tandem colonoscopy

INTERVENTIONS:
Diagnostic Test: Tandem colonoscopy — Different image enhanced endoscopy systems

SUMMARY:
This is a prospective randomized trial comparing the adenoma detection rate of LCI with NBI. Eligible patients are randomly allocated in a 1:1 ratio to undergo tandem colonoscopy with LCI (LCI group) or NBI (NBI group). Randomization will be carried out by computer generated random sequences and stratified according to endoscopist's experiences (experienced versus fellows) and indications of colonoscopy (symptomatic vs screening/surveillance).

The primary outcome of this study is to compare the adenoma or polyp detection rates by LCI and NBI during the first examination. Secondary outcomes included adenoma/polyp miss rate by LCI or NBI. Other outcomes include sessile serrated adenomas or polyps (SSA/P) detection rates and advanced adenoma detection rates.

DETAILED DESCRIPTION:
Study design and randomization:

This is a prospective randomized head-to-head trial comparing the adenoma detection rate of LCI with NBI. Eligible patients are randomly allocated in a 1:1 ratio to undergo tandem colonoscopy with LCI (LCI group) or NBI (NBI group). Randomization will be carried out by computer generated random sequences and stratified according to endoscopist's experiences (experienced versus fellows) and indications of colonoscopy (symptomatic vs screening/surveillance). All procedures are performed with high-definition endoscopes and the LASEREO endoscopic system (Fujifilm Co, Tokyo, Japan) or the EVIS- EXERA 290 video system (Olympus Optical, Tokyo, Japan).

Colonoscopy:

Patients are instructed to take low-residue diet two days before colonoscopy. Oral polyethylene glycol lavage solution is used for bowel preparation (routine bowel preparation). The assigned endoscopic system will be used and the colonoscope will advance to cecum under WL in all patients. Cecal intubation is confirmed by identification of the appendiceal orifice and ileocecal valve or by intubation of the ileum. Once cecal intubation is performed, the colonoscope is withdrawn to the anus under LCI or NBI accordingly. All detected polyps will be removed during this examination. The withdrawal time of the first pass (minus the polypectomy site) will be measured by a stopwatch.

The size (measured with biopsy forceps), location, and morphology of polyps are recorded by an independent observer. The Boston Bowel Preparation Scale score is evaluated during examination.

Immediately after the first pass examination, a second examination will be performed by the same colonoscope and the same endoscopist. The colonoscope will be reintroduced to the cecum using WL and withdraw using the previously assigned method (ie LCI or NBI). Any polyp detected on second pass examination will be removed and the withdrawal time of the second pass will also be documented. All polyp specimens are clearly labelled for histological examination.

Histologic examination All resected and biopsy specimens are fixed in 10% buffered formalin solution, and examined histologically by hematoxylin and eosin staining. The histopathological diagnosis is determined by experienced pathologists, who are blinded to the assigned endoscopic system, according to the World Health Organization (WHO) criteria.Advanced adenomas are defined as adenoma ≥10 mm in diameter or with villous histology in 25% or high-grade dysplasia (HGD), or carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients undergoing outpatient colonoscopy
* aged 40 or above

Exclusion Criteria:

* unable to provide informed consent
* have undergone previous colorectal resection
* personal history of colorectal cancer, inflammatory bowel disease, familial adenomatous polyposis, Peutz-Jeghers syndrome, or other polyposis syndromes
* considered to be unsafe for polypectomy including patients with bleeding tendency and those with severe comorbid illnesses
* cecum could not be intubated for various reasons or due to poor bowel preparation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma/polyp detection rate | first-pass colonoscopy
  Percentage of patients with adenoma/polyp detected

SECONDARY OUTCOMES:
Adenoma/polyp miss rate | second-pass colonoscopy
  percentage of patients with adenoma/polyp missed

OTHER OUTCOMES:
advanced adenoma detection rate | first-pass colonoscopy
  percentage of patients with advanced adenoma
SSA detection rate | first-pass colonoscopy
  percentage of patients with sessile serrated adenoma/polyp

CONTACTS AND LOCATIONS:
Overall Officials: Wai K Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung WK, Guo CG, Ko MKL, To EWP, Mak LY, Tong TSM, Chen LJ, But DYK, Wong SY, Liu KSH, Tsui V, Lam FYF, Lui TKL, Cheung KS, Lo SH, Hung IFN. Linked color imaging versus narrow-band imaging for colorectal polyp detection: a prospective randomized tandem colonoscopy study. Gastrointest Endosc. 2020 Jan;91(1):104-112.e5. doi: 10.1016/j.gie.2019.06.031. Epub 2019 Jul 2. PMID 31276672